CLINICAL TRIAL: NCT04898816
Title: Comparing the Effectiveness of Cyanoacrylate Tissue Adhesives and Conventional Sutures in the Closure of Intraoral Surgical Wounds- A Randomized Clinical Trial
Brief Title: Comparing the Effectiveness of Cyanoacrylate Tissue Adhesives and Conventional Sutures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Abdul Kalam Azad, Assistant Professor, Melaka Manipal Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMMC/FOD/AR/B8/E C-2020 (08)
Record Dates: First submitted 2021-04-28; First posted 2021-05-24 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Application of cyanoacrylate tissue adhesive over the surgical wound
  Interventions: Procedure: closure of wound using n- butyl 2-octyl cyanoacrylate tissue adhesive
- Group B (Active Comparator): Suturing the surgical wound using braided black silk
  Interventions: Procedure: closure of wound using braided silk suture

INTERVENTIONS:
Procedure: closure of wound using n- butyl 2-octyl cyanoacrylate tissue adhesive — Application of cyanoacrylate tissue adhesives over the surgical wound
  Arms: Group A
Procedure: closure of wound using braided silk suture — suturing the surgical wound using braided black silk
  Arms: Group B

SUMMARY:
This study compares the effectiveness of two materials used for intraoral wound closure after removal of impacted mandibular third molar tooth. One Group received braided black silk suture and the other group received N-butyl 2-octyl cyanoacrylate tissue adhesives.

DETAILED DESCRIPTION:
Conventional method of wound closure after removal of impacted mandibular molar is by suturing the wound using braided black silk suture and allowing for primary healing. Suturing in the most posterior region of oral cavity is not easy, it requires more time and additional skills as well. Patient has to come for a second visit for removal of suture. Moreover tight sutures may lead to ischemia and necrosis.

Tissue adhesives adopts the idea of sutureless wound closure. They are even sloughed off from the surface of mucosa 7 days after the application.

This study compares the effectiveness of conventional sutures and tissue adhesives in closure of intraoral surgical wounds after removal of mandibular third molar.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring surgical removal of mesioangular, position A impacted mandibular third molar
* clean incisions approximately 2-3 cms in length which can be approximated
* Healthy (ASAI) or patients with mild systemic disease no functional limitations
* Patients not allergic to the drugs or anesthetic agents used in the surgical protocol

Exclusion Criteria:

* Patients taking any medications that influences wound healing
* Patients on non steroidal anti inflammatory drugs
* smokers
* uncooperative patients patients allergic to cyanoacrylate

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 1st postoperative day
  A 10 mm Numerical rating scale assessing postoperative pain. Possible score ranges from 0 (no pain) to 10 (worst possible pain).
postoperative pain | 2nd postoperative day
  A 10 mm Numerical rating scale assessing postoperative pain. Possible score ranges from 0 (no pain) to 10 (worst possible pain).
Postoperative pain | 3rd postoperative day
  A 10 mm Numerical rating scale assessing postoperative pain. Possible score ranges from 0 (no pain) to 10 (worst possible pain).
Postoperative pain | 4th postoperative day
  A 10 mm Numerical rating scale assessing postoperative pain. Possible score ranges from 0 (no pain) to 10 (worst possible pain).
postoperative pain | 5th postoperative day
  A 10 mm Numerical rating scale assessing postoperative pain. Possible score ranges from 0 (no pain) to 10 (worst possible pain).
wound healing | 7th postoperative day
  A 5 point early wound healing scale assessing wound healing after 7 postoperative days.

CONTACTS AND LOCATIONS:
Overall Officials: abdul K azad, Principal Investigator — Melaka Manipal Medical College
Locations (1):
- Melaka Manipal Medical College, Melaka Tengah, Melaka, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 month
Access Criteria: Study protocol will be provided only if requested through a proper channel, dean of college , with proper justification.